CLINICAL TRIAL: NCT03973931
Title: Personalized Patient Data and Behavioral Nudges to Improve Adherence to Chronic Cardiovascular Medications (The Nudge Study)
Brief Title: Personalized Patient Data and Behavioral Nudges to Improve Adherence to Chronic Cardiovascular Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-2779; UH3HL144163 (NIH)
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases; Adherence, Medication; Medication Adherence; Diabetes Mellitus; Hypertension; Hyperlipidemias; Coronary Artery Disease; Atrial Fibrillation
Keywords: cardiovascular disease; telemedicine; medication adherence; behavioral health
MeSH Terms: conditions — Cardiovascular Diseases; Medication Adherence; Diabetes Mellitus; Hypertension; Hyperlipidemias; Coronary Artery Disease; Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: The study will be a pragmatic, randomized controlled study with four treatment arms. Once patients are identified through pharmacy refill data to have a 7-day gap in any prescribed CV medication refills, they will be randomized to one of four arms, described in Intervention below. Randomization will be stratified within each of the clinics, and within strata defined by number of other CV medication classes that are prescribed at randomization (1-4), using blocks of 4 patients to ensure balance within clinics over time. Thus, within each clinic and number of other medication stratum, each set of 4 consecutively enrolled subjects will be randomized to the four study arms. Treatments will be initiated immediately upon randomization, in response to the 7-day gap.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual Care (No Intervention): This group will not receive an intervention. We have included a usual care group to demonstrate the impact of the text messaging interventions above and beyond usual care given that many prior medication adherence interventions have demonstrated small to negligible effects.
- Generic Nudge (Experimental): A generic reminder text will be delivered to patients to refill their medication at days 1, 3, 5, 7 and 10 after they been labeled as non-adherent.
  Interventions: Behavioral: Nudge
- Optimized nudge (Experimental): An optimized nudge text will be delivered to patients to remind them to refill their medications at days 1, 3, 5, 7 and 10 after they have been labeled as non-adherent.
  Interventions: Behavioral: Nudge
- Optimized nudge plus AI Chat Bot (Experimental): An optimized nudge text will be delivered to patients to remind them to refill their medications at days 1 and 3 after they have been labeled as non-adherent. If the patient has not filled their medication on days 5 and 7, in addition to receiving an optimized nudge text, an AI will conduct interactive chat via a chat bot to assess barriers filling the medication as described in Aim 1 above. If they still have not filled the medication, they will receive another message on day 10.
  Interventions: Behavioral: Nudge

INTERVENTIONS:
Behavioral: Nudge — Interventions will include a variety of text messages aimed at improving medication adherence.
  Arms: Generic Nudge; Optimized nudge; Optimized nudge plus AI Chat Bot

SUMMARY:
The study plans to learn if sending different text messages, serving as reminders or encouragement, may help patients take their medication more often if they have had trouble keeping up with their medicines.

DETAILED DESCRIPTION:
Background: Up to fifty percent of patients do not take their cardiovascular medications as prescribed resulting in increased morbidity, mortality, and healthcare costs. Mobile and digital technologies for health promotion and disease self-management offer an intriguing and as of yet untested opportunity to adapt behavioral 'nudges' using ubiquitous cell phone technology to facilitate medication adherence.

Objectives: Aim 1: Conduct a pragmatic patient-level randomized intervention across three health care systems (HCS) to improve adherence to chronic CV medications. The primary outcome will be medication adherence defined by the proportion of days covered (PDC) using pharmacy refill data. Secondary outcomes include clinical events (e.g., event times for stroke, MI, mortality), utilization of care (e.g., hospitalizations or clinic visits for CV-related reasons), and costs of healthcare utilization. Aim 2: Evaluate the intervention using a mixed methods approach and applying the RE-AIM (reach, effectiveness, adoption, implementation, and maintenance) framework. In addition, assess the context and implementation processes to inform local tailoring, adaptations and modifications, and eventual expansion of the intervention within the 3 HCS more broadly and nationally.

Setting: The study will be conducted within three HCS in metro Denver: VA Eastern Colorado Health Care System (VA), Denver Health and Hospital Authority, and UCHealth.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following cardiovascular conditions and respective medication classes:
* Hypertension (Beta-blockers [B-blockers)], Calcium Channel Blocker [CCB], Angiotensin converting enzyme inhibitors (ACEi), Angiotensin Receptor Blockers [ARB], or Thiazide diuretic)
* Hyperlipidemia (HMG CoA reductase inhibitor [Statins])
* Diabetes (Alpha-glucosidase inhibitors, Biguanides, DPP-4 inhibitors, Sodium glucose transport inhibitor, Meglitinides, Sulfonylureas, Thiazolidinediones, or statins Coronary artery disease P2Y12 inhibitor [Clopidogrel, Ticagrelor, Prasugrel, Ticlopidine], B-blockers, ACEi or ARB or statins)
* Atrial fibrillation (Direct oral anticoagulants, B-blockers, CCB)

Exclusion Criteria:

* Patients who do not have a mailing address listed in EHR;
* Patients who do not have a landline or cellphone listed in EHR;
* Currently pregnant if denoted in the EHR at the time of the data pull;
* Patients with a mailing address outside of the state of Colorado;
* Patients that do not speak either English or Spanish.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9501 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ho, MD, PhD, Principal Investigator — University of Colorado, Denver; Sheana Bull, PhD, MPH, Principal Investigator — University of Colorado, Denver
Locations (4):
- United States (4):
  - UCHealth, Aurora, Colorado
  - University of Colorado Denver, Aurora, Colorado
  - VA Eastern Colorado Health Care System, Aurora, Colorado
  - Denver Health and Hospital Authority, Denver, Colorado

IPD SHARING:
Plan to Share IPD: Yes
Data collected as part of this project will be released in accordance with standard data sharing policies and procedures. Data will be made available to the broader scientific community after results are published in peer-reviewed journals.
  Prior to making this data available, data will be redacted to strip identifiers and further de-identified by removing indirect identifiers that could lead to "deductive disclosure" of identities.
  Due to the small numbers of participants in the qualitative interviews, we do not anticipate sharing raw data from individuals.
  The agreement will prohibit the recipient from transferring the data to other users, require that the data's security be protected by standard means and be used for research purposes only. After a requestor completes the data-sharing agreement, we will either mail a CD with a limited dataset to the requestor, or email the data through our secure email system that requires users to create an account to receive sensitive data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be shared in a timely manner, as requested.
Access Criteria: The study team will share technical and practical knowledge regarding the creation of the chat bot and text messaging intervention, upon request. Further, the study team would readily share all data collection instruments and assessment algorithms used in the project to qualified individuals within the scientific community with the agreement that they will appropriately acknowledge the study team who developed the instruments.

REFERENCES:
- [Background] Jackevicius CA, Li P, Tu JV. Prevalence, predictors, and outcomes of primary nonadherence after acute myocardial infarction. Circulation. 2008 Feb 26;117(8):1028-36. doi: 10.1161/CIRCULATIONAHA.107.706820. PMID 18299512
- [Background] Ho PM, Spertus JA, Masoudi FA, Reid KJ, Peterson ED, Magid DJ, Krumholz HM, Rumsfeld JS. Impact of medication therapy discontinuation on mortality after myocardial infarction. Arch Intern Med. 2006 Sep 25;166(17):1842-7. doi: 10.1001/archinte.166.17.1842. PMID 17000940
- [Background] Rasmussen JN, Chong A, Alter DA. Relationship between adherence to evidence-based pharmacotherapy and long-term mortality after acute myocardial infarction. JAMA. 2007 Jan 10;297(2):177-86. doi: 10.1001/jama.297.2.177. PMID 17213401
- [Background] Spertus JA, Kettelkamp R, Vance C, Decker C, Jones PG, Rumsfeld JS, Messenger JC, Khanal S, Peterson ED, Bach RG, Krumholz HM, Cohen DJ. Prevalence, predictors, and outcomes of premature discontinuation of thienopyridine therapy after drug-eluting stent placement: results from the PREMIER registry. Circulation. 2006 Jun 20;113(24):2803-9. doi: 10.1161/CIRCULATIONAHA.106.618066. Epub 2006 Jun 12. PMID 16769908
- [Background] Brown MT, Bussell JK. Medication adherence: WHO cares? Mayo Clin Proc. 2011 Apr;86(4):304-14. doi: 10.4065/mcp.2010.0575. Epub 2011 Mar 9. PMID 21389250
- [Background] Wei L, Wang J, Thompson P, Wong S, Struthers AD, MacDonald TM. Adherence to statin treatment and readmission of patients after myocardial infarction: a six year follow up study. Heart. 2002 Sep;88(3):229-33. doi: 10.1136/heart.88.3.229. PMID 12181210
- [Background] Wei L, Flynn R, Murray GD, MacDonald TM. Use and adherence to beta-blockers for secondary prevention of myocardial infarction: who is not getting the treatment? Pharmacoepidemiol Drug Saf. 2004 Nov;13(11):761-6. doi: 10.1002/pds.963. PMID 15386713
- [Background] Lu CY, Ross-Degnan D, Soumerai SB, Pearson SA. Interventions designed to improve the quality and efficiency of medication use in managed care: a critical review of the literature - 2001-2007. BMC Health Serv Res. 2008 Apr 7;8:75. doi: 10.1186/1472-6963-8-75. PMID 18394200
- [Background] Volpp KG, Loewenstein G, Troxel AB, Doshi J, Price M, Laskin M, Kimmel SE. A test of financial incentives to improve warfarin adherence. BMC Health Serv Res. 2008 Dec 23;8:272. doi: 10.1186/1472-6963-8-272. PMID 19102784
- [Background] Murray MD, Young J, Hoke S, Tu W, Weiner M, Morrow D, Stroupe KT, Wu J, Clark D, Smith F, Gradus-Pizlo I, Weinberger M, Brater DC. Pharmacist intervention to improve medication adherence in heart failure: a randomized trial. Ann Intern Med. 2007 May 15;146(10):714-25. doi: 10.7326/0003-4819-146-10-200705150-00005. PMID 17502632
- [Background] Lee JK, Grace KA, Taylor AJ. Effect of a pharmacy care program on medication adherence and persistence, blood pressure, and low-density lipoprotein cholesterol: a randomized controlled trial. JAMA. 2006 Dec 6;296(21):2563-71. doi: 10.1001/jama.296.21.joc60162. Epub 2006 Nov 13. PMID 17101639
- [Background] Peterson PN, Campagna EJ, Maravi M, Allen LA, Bull S, Steiner JF, Havranek EP, Dickinson LM, Masoudi FA. Acculturation and outcomes among patients with heart failure. Circ Heart Fail. 2012 Mar 1;5(2):160-6. doi: 10.1161/CIRCHEARTFAILURE.111.963561. Epub 2012 Jan 13. PMID 22247483
- [Background] Gurol-Urganci I, de Jongh T, Vodopivec-Jamsek V, Atun R, Car J. Mobile phone messaging reminders for attendance at healthcare appointments. Cochrane Database Syst Rev. 2013 Dec 5;2013(12):CD007458. doi: 10.1002/14651858.CD007458.pub3. PMID 24310741
- [Background] de Jongh T, Gurol-Urganci I, Vodopivec-Jamsek V, Car J, Atun R. Mobile phone messaging for facilitating self-management of long-term illnesses. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD007459. doi: 10.1002/14651858.CD007459.pub2. PMID 23235644
- [Background] Vodopivec-Jamsek V, de Jongh T, Gurol-Urganci I, Atun R, Car J. Mobile phone messaging for preventive health care. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD007457. doi: 10.1002/14651858.CD007457.pub2. PMID 23235643
- [Derived] Ho PM, Glorioso TJ, Allen LA, Blankenhorn R, Glasgow RE, Grunwald GK, Khanna A, Magid DJ, Marrs JC, Novins-Montague S, Orlando S, Peterson P, Plomondon ME, Sandy LM, Saseen JJ, Trinkley KE, Vaughn S, Waughtal J, Bull S. Personalized Patient Data and Behavioral Nudges to Improve Adherence to Chronic Cardiovascular Medications: A Randomized Pragmatic Trial. JAMA. 2025 Jan 7;333(1):49-59. doi: 10.1001/jama.2024.21739. PMID 39621340
- [Derived] Glasgow RE, Knoepke CE, Magid D, Grunwald GK, Glorioso TJ, Waughtal J, Marrs JC, Bull S, Ho PM. The NUDGE trial pragmatic trial to enhance cardiovascular medication adherence: study protocol for a randomized controlled trial. Trials. 2021 Aug 11;22(1):528. doi: 10.1186/s13063-021-05453-9. PMID 34380527
- [Derived] Luong P, Glorioso TJ, Grunwald GK, Peterson P, Allen LA, Khanna A, Waughtal J, Sandy L, Ho PM, Bull S. Text Message Medication Adherence Reminders Automated and Delivered at Scale Across Two Institutions: Testing the Nudge System: Pilot Study. Circ Cardiovasc Qual Outcomes. 2021 May;14(5):e007015. doi: 10.1161/CIRCOUTCOMES.120.007015. Epub 2021 May 17. PMID 33993727
- See also: NIH Collaboratory Site discussing the Nudge Project — https://rethinkingclinicaltrials.org/demonstration-projects/ug3-project-personalized-patient-data-and-behavioral-nudges-to-improve-adherence-to-chronic-cardiovascular-medications-nudge/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Generic Nudge | Optimized Nudge | Optimized Nudge Plus AI Chat Bot | Usual Care
Started | 2377 | 2373 | 2375 | 2376
Completed | 2324 | 2305 | 2319 | 2321
Not Completed | 53 | 68 | 56 | 55
Not completed — Lost to Follow-up | 47 | 63 | 51 | 54
Not completed — opted out | 6 | 5 | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Generic Nudge | Optimized Nudge | Optimized Nudge Plus AI Chat Bot | Usual Care | Total
Number analyzed (Participants) | 2324 | 2305 | 2319 | 2321 | 9269
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (12.5) | 60 (12.9) | 60.1 (12.7) | 60.1 (12.6) | 60.0 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1087 | 1075 | 1101 | 1088 | 4351
  Male | 1237 | 1230 | 1218 | 1233 | 4918
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1100 | 1147 | 1168 | 1149 | 4564
  Not Hispanic or Latino | 1204 | 1141 | 1134 | 1150 | 4629
  Unknown or Not Reported | 20 | 17 | 17 | 22 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 22 | 27 | 23 | 35 | 107
  Asian | 29 | 31 | 21 | 29 | 110
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 6 | 3 | 14
  Black or African American | 391 | 378 | 356 | 392 | 1517
  White | 1601 | 1615 | 1646 | 1598 | 6460
  More than one race | 10 | 14 | 16 | 9 | 49
  Unknown or Not Reported | 268 | 238 | 251 | 255 | 1012
Marital Status [Count of Participants; unit: Participants]
  Married Married | 994 | 940 | 980 | 950 | 3864
  Single | 883 | 883 | 870 | 874 | 3510
  Divorced/Widowed | 434 | 464 | 452 | 483 | 1833
  Unknown | 13 | 18 | 17 | 14 | 62
Insurance [Count of Participants; unit: Participants]
  Medicare | 853 | 878 | 860 | 889 | 3480
  Medicaid | 659 | 632 | 629 | 665 | 2585
  Commercial | 463 | 471 | 500 | 441 | 1875
  Unknown | 123 | 96 | 130 | 112 | 461
  VHA | 8 | 7 | 8 | 12 | 35
  None | 218 | 221 | 192 | 202 | 833
Medical History [Number; unit: participants]
  Depression | 421 | 463 | 442 | 416 | 1742
  Chronic Kidney Disease | 191 | 202 | 203 | 189 | 785
  Heart Failure | 160 | 199 | 163 | 171 | 693
  Cerebrovascular Disease | 142 | 145 | 125 | 134 | 546
  Posttraumatic Stress Disorder | 118 | 114 | 102 | 108 | 442
  Substance Abuse | 89 | 101 | 116 | 88 | 394
  Prior Coronary Revascularization | 63 | 56 | 70 | 58 | 247
  Prior Myocardial Infarction | 95 | 109 | 121 | 98 | 423
Qualifying Condition [Number; unit: participants]
  Hypertension | 1837 | 1829 | 1821 | 1864 | 7351
  Diabetes | 1148 | 1164 | 1162 | 1149 | 4623
  Hyperlipidemia | 1072 | 1052 | 1089 | 1054 | 4267
  Coronary Artery Disease | 305 | 325 | 352 | 328 | 1310
  Atrial Fibrillation | 132 | 152 | 130 | 134 | 548
  >1 Qualifying Condition | 1406 | 1390 | 1410 | 1438 | 5644
Baseline Medication Classes [Count of Participants; unit: Participants]
  1 Active Class | 597 | 564 | 567 | 557 | 2285
  2 Active Classes | 551 | 572 | 584 | 591 | 2298
  >=3 Active Classes | 1176 | 1169 | 1168 | 1173 | 4686
Intervention Delivery [Count of Participants; unit: Participants]
  Text Messages | 2126 | 2089 | 2117 | 0 | 6332
  Interactive Voice Response Telephone Messages | 198 | 216 | 202 | 0 | 616
  No Text or IVR | 0 | 0 | 0 | 2321 | 2321

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence
Description: The primary outcome was medication adherence defined by the proportion of days covered (PDC) using pharmacy refill data adjusted difference from usual care.
Time Frame: 12 months after intervention
Population: mean pdc at 12 months
Measure: Mean (95% Confidence Interval); unit: mean PDC
Arm/Group | Generic Nudge | Optimized Nudge | Optimized Nudge Plus AI Chat Bot | Usual Care
Number analyzed (Participants) | 2324 | 2305 | 2319 | 2321
mean PDC | .606 [.594 to .618] | .620 [.609 to .633] | .623 [.612 to .635] | .630 [.618 to .640]
Statistical Analysis 1: Comparison: Generic Nudge vs Optimized Nudge vs Optimized Nudge Plus AI Chat Bot vs Usual Care; Test type: Non-Inferiority — Generalized Estimating Equation (GEE) model with an identity link and independence with unequal variances for the covariance structure of the 12 observations; p < 0.05, GEE; To account for multiple treatment comparisons significance levels of 0.05/3

2. Primary Outcome: Mean Proportion of Days Covered Relative to Usual Care
Description: We analyzed this longitudinal data (up to 12 observations per patient) and estimated absolute differences in PDC between treatment arms and usual care using a Generalized Estimating Equation (GEE) model with an identity link and independence with unequal variances for the covariance structure of the 12 observations .A multistage gatekeeper approach was used to account for multiple treatment comparisons by comparing each of the 3 treatment arms to the control in stage 1 using significance levels of 0.05/3, and if any test was significant, a significance level of (R/3)*(0.05/3) using the Holm method was used for the 3 pairwise comparisons, where R is the number of significant stage 1 tests.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: proportion of days covered
Arm/Group | Generic Nudge | Optimized Nudge | Optimized Nudge Plus AI Chat Bot
Number analyzed (Participants) | 2324 | 2305 | 2319
proportion of days covered | 0.022 [0.003 to 0.042] | 0.020 [0.001 to 0.039] | 0.023 [0.004 to 0.042]
Statistical Analysis 1: Comparison: Generic Nudge vs Optimized Nudge vs Optimized Nudge Plus AI Chat Bot; Test type: Non-Inferiority — Analysis of the longitudinal data (12 observations per patient) and estimated absolute differences in PDC between treatment group and usual care was analyzed using Generalized Estimating Equation (GEE) model with an identity link and independence with unequal variances for the covariance structure was used; p < 0.05, GEE — To account for multiple treatment comparisons significance levels of 0.05/3, and if any test was significant, a significance level of (R/3)*(0.05/3) using the Holm method was used for the 3 pairwise comparisons, R=number of significant stage 1 tests

3. Secondary Outcome: Hospitalization
Description: estimated probability of hospitalization at one year
Time Frame: one year
Population: 1-year Kaplan-Meier rate estimates with 95% confidence intervals.
Measure: Mean (95% Confidence Interval); unit: estimated probability of hospitalization
Arm/Group | Generic Nudge | Optimized Nudge | Optimized Nudge Plus AI Chat Bot | Usual Care
Number analyzed (Participants) | 2324 | 2305 | 2319 | 2321
estimated probability of hospitalization | .13 [.115 to .144] | .136 [.121 to .151] | .136 [.121 to .151] | .143 [.128 to .158]

4. Secondary Outcome: Death
Description: estimated probability of death at one year
Time Frame: one year
Population: 1-year Kaplan-Meier rate estimates with 95% confidence intervals.
Measure: Mean (95% Confidence Interval); unit: estimated probability of death
Arm/Group | Generic Nudge | Optimized Nudge | Optimized Nudge Plus AI Chat Bot | Usual Care
Number analyzed (Participants) | 2324 | 2305 | 2319 | 2321
estimated probability of death | .031 [.03 to .039] | .026 [.019 to .033] | .027 [.020 to .034] | .033 [.025 to .041]

5. Secondary Outcome: Emergency Department Visit
Description: estimated probability of emergency department visit at one year
Time Frame: one year
Population: 1-year Kaplan-Meier rate estimates with 95% confidence intervals.
Measure: Mean (95% Confidence Interval); unit: estimated probability of ED visit
Arm/Group | Generic Nudge | Optimized Nudge | Optimized Nudge Plus AI Chat Bot | Usual Care
Number analyzed (Participants) | 2324 | 2305 | 2319 | 2321
estimated probability of ED visit | .292 [.272 to .311] | .285 [.265 to .305] | .294 [.274 to .313] | .301 [.281 to .321]

ADVERSE EVENTS:
Time Frame: 12 months
Description: All-Cause Mortality
Arm/Group | Generic Nudge | Optimized Nudge | Optimized Nudge Plus AI Chat Bot | Usual Care
All-Cause Mortality (participants affected / at risk) | 63/2324 | 53/2305 | 55/2319 | 68/2321
Serious Adverse Events (participants affected / at risk) | 267/2324 | 283/2305 | 283/2319 | 303/2321
Other Adverse Events (participants affected / at risk) | 612/2324 | 594/2305 | 616/2319 | 639/2321
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Generic Nudge (N=2324) | Optimized Nudge (N=2305) | Optimized Nudge Plus AI Chat Bot (N=2319) | Usual Care (N=2321)
Number with All Cause Hospitalization in 12 months (General disorders) | 267 (267) | 283 (283) | 283 (283) | 303 (303) — Number of participants with all cause hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Generic Nudge (N=2324) | Optimized Nudge (N=2305) | Optimized Nudge Plus AI Chat Bot (N=2319) | Usual Care (N=2321)
Number with Emergency Department visits in 12 months (General disorders) | 612 (612) | 594 (594) | 616 (616) | 639 (639) — Number of participants with all cause ED visits at12 months

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT03973931/Prot_SAP_000.pdf